CLINICAL TRIAL: NCT01827813
Title: Comparison Of Effectiveness of Transrectal Ultrasonography-Guided Saturation Biopsy And 10-12 Core Biopsy In Repeated Prostate Biopsies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Abdullah Demirtas, Assistant Professor, TC Erciyes University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ProstatBX
Record Dates: First submitted 2013-04-01; First posted 2013-04-10 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Cancer
Keywords: prostate-specific antigen; digital rectal examination; transrectal ultrasonography; needle biopsy; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saturation biopsy (Active Comparator): Saturation biopsy was performed in left lateral decubitus position after application of sedo-analgesia by the anesthesiologists on an outpatient basis. After preparation of the rectal ultrasound probe and assuming an appropriate position, ultrasonographic examination of the prostate was performed on axial and sagittal plane. After injecting 3 cc of prilocaine to each of the right and left lobes in the right and left periprostatic region, prostatic size was measured and changes in the zonal anatomy and ultrasonographic view of the tissue were defined. Next, biopsy procedure was performed with an 18 G, 20 cm tru-cut biopsy needle and an automatic biopsy gun. After passing beyond the rectal mucosa, the needle was advanced until 0.5 cm proximal to the area of interest by tracking the image of the needle on the screen. As a total,24,26 or 28 biopsies were taken depending on prostate volume.
  Interventions: Procedure: Transrectal prostate biopsy with ultrasonography.; Procedure: Periprostatic block; Procedure: Sedoanalgesia
- 10-12 core biopsy (Active Comparator): 10-12 core biopsy was performed in left lateral decubitus position without sedo-analgesia on an outpatient basis. After preparation of the probe and assuming an appropriate position, ultrasonographic examination of the prostate was performed on axial and sagittal plane. After injecting 3 cc of prilocaine to each of the right and left lobes in the right and left periprostatic region, prostatic size was measured and changes in the zonal anatomy and ultrasonographic view of the tissue were defined. Next, biopsy procedure was performed with an 18 G, 20 cm tru-cut biopsy needle and an automatic biopsy gun. As a total 10 or 12 core biopsies were taken depending on prostate volume. The biopsies were taken form right base, right mid, right apex, right far-lateral base, right far-lateral mid and left base, left apex, left far-lateral base, and left far-lateral mid in 10 core biopsy, also two additional transitional zone biopsies were taken in 12 core biopsies.
  Interventions: Procedure: Transrectal prostate biopsy with ultrasonography.; Procedure: Periprostatic block

INTERVENTIONS:
Procedure: Transrectal prostate biopsy with ultrasonography. — Transrectal prostate biopsy was performed in left lateral decubitus position with sedo-analgesia in saturation biopsy group and without sedoanalgesia in 10-12 core biopsy group on outpatient basis. After preparation of the rectal ultrasound probe and assuming an appropriate position, ultrasonographic examination of the prostate was performed on axial and sagittal plane. Periprostatic block was performed with the injection of 3 cc of prilocaine to each of the right and left lobes in the right and left periprostatic region in both groups before biopsy. Biopsy procedure was performed with an 18 G, 20 cm tru-cut biopsy needle and an automatic biopsy gun. After passing beyond the rectal mucosa, the needle was advanced until 0.5 cm proximal to the area of interest by tracking the image of the needle on the screen.
Procedure: Periprostatic block — Periprostatic block was used for local anesthesia. 3 cc 2% prilocaine was injected to both periprostatic region in both saturation biopsy and 10-12 core biopsy group with transrectal ultrasonography.
Procedure: Sedoanalgesia — Sedoanalgesia was used in saturation biopsy group. It was given by an anesthesiologist. Patients were given adequate counselling regarding sedoanesthesia as well as the biopsy procedure. They were advised to fast the night before the procedure.Before induction of sedoanalgesia all patients were monitorized for peripheric oxygen saturation and electrocardiography (ECG).Additionally nasal oxygen with 3ml/min was given to all patients by nasal canula.Sedoanalgesia was induced with 0.05mg/kg of midazolam, 1mg/kg of propofol and 1mg/kg of fentanyl. additional propofol was given with dose of 0.3mg/kg as patients needed.
  Arms: Saturation biopsy

SUMMARY:
OBJECTIVE To assessment the results of repeated saturation and 10-12 core biopsy protocols in patients with a negative initial biopsy but continued suspicion for prostate cancer MATERIALS AND METHOD Data of the patients who underwent prostate biopsy between June 2007 and June 2012 were retrospectively assessed. Patients with an abnormal digital examination findings and/or abnormal serum prostate specific antigen levels were biopsied. The indication for a repeated biopsy was determined as the continued suspicion for a malignancy after the initial benign biopsy result and/or a pathology result consistent with a high-grade prostatic intraepithelial neoplasia or atypical small acinar proliferation. Patients who underwent saturation and core 10-12 biopsies at repeated biopsies were compared. Statistical analyses were performed with Shapiro-Wilk test and Mann- Whitney U test. A p value less than 0.05 was accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Abnormal digital examination
2. High serum prostate specific antigen (PSA) level.
3. The continued suspicion for a malignancy after the initial benign biopsy result and/or a pathology result consistent with a high-grade prostatic intraepithelial neoplasia (HGPIN) or atypical small acinar proliferation (ASAP).

Exclusion Criteria:

1. Patients with coagulopathies
2. Patients with unsuitable general conditions for prostate biopsy.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-06; Primary Completion 2012-06 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Detection rate of prostate cancer. | At least two months
  Prostate cancer detection rate after saturation and repeated 10-12 core prostate biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Demirtas, Assistant Prof., MD, Study Director — Erciyes University, Faculty of Medicine; Akın Avcı, Resident in UrologyMD,, Principal Investigator — Erciyes University, Faculty of Medicine; Ibrahim Gulmez, Professor in Urology,M.D., Study Chair — Erciyes University, Faculty of Medicine
Locations (1):
- Department of Urology, Ercieys University, Faculty Of Medicine,, Kayseri, Turkey (Türkiye)